CLINICAL TRIAL: NCT04459416
Title: Opioid-Sparing Pain Treatment In Myeloma And Lymphoma Patients Undergoing High-Dose Chemotherapy (OPTIMAL-HiChemo): Randomized Controlled Trial
Brief Title: Managing Pain and Symptom Burden Caused by Chemotherapy in People With Myeloma or Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-264
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma; Hodgkin Disease; Non-Hodgkin Lymphoma
Keywords: Pain management; Acupuncture; 20-264
MeSH Terms: conditions — Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Agnosia | interventions — Acupuncture Therapy; Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: This is a multicenter, two-arm randomized controlled trial. Randomization will be stratified by study site, primary cancer diagnosis (MM versus HD versus NHL) and transplantation setting (inpatient versus outpatient) to ensure these characteristics are comparably distributed between the two study arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care plus Acupuncture (Experimental): Acupuncture will start on Day 0 and continue once daily to Day 15, as long as the patient is inpatient or comes to the clinic for post-transplantation follow-up. to prevent severe pain. If acupuncture does not prevent severe pain, the participant will receive opioid medication as backup pain relief.
  Interventions: Other: Acupuncture; Drug: opioid; Other: Assessments
- Usual Care (Active Comparator): Will receive only the usual pain management approach, which includes opioid medication when needed for severe pain, according to the routine guidelines for their care.
  Interventions: Drug: opioid; Other: Assessments

INTERVENTIONS:
Other: Acupuncture — Acupuncture treatments will be scheduled to cover the period of high symptom burden. Acupuncture will start on Day 0 and continue once daily to Day 15, as long as the patient is inpatient or comes to the clinic for post-transplantation follow-up. Electrical stimulation (e-acupuncture) may be applied to the ST36 and SP6 points when appropriate as per standard acupuncture practice.
  Arms: Usual Care plus Acupuncture
Drug: opioid — All study patients will receive the usual HSCT care and pain management regimens (usually opioids) as per standard practice at the study institution.
Other: Assessments — Participants will be asked to complete patient reported outcomes assessments online using REDCap or, If they prefer, via pencil and paper or over the phone. Assessments at baseline (within 4 weeks before HiChemo) and on or about days 7, 15, 30, and 90 after the first dose of HiChemo.

SUMMARY:
The purpose of this study is to find out whether acupuncture treatments can reduce the need for opioid medication when managing pain caused by chemotherapy. The study will compare the effects of adding acupuncture to usual pain management with those of usual pain management alone, in reducing opioid use by relieving pain. Researchers also want to find out more about the effects of acupuncture treatments on other symptoms caused by cancer treatments and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* pathological diagnosis of MM, HD or NHL
* scheduled for high dose chemotherapy for auto-HSCT in the following month (30 days)
* not taking opioids regularly in the week prior to consent (one-time dosing of opioids for a painful procedure is allowed)

Exclusion Criteria:

* absolute neutrophil count (ANC) of <500/μl, platelet count of <20,000/ μl or INR >2.0
* acupuncture within two weeks prior to HiChemo (to avoid residual effects of acupuncture)
* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jun Mao, MD, MSCE, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancel Care Alliance (Data Collection Only), Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture Plus Usual Care: Acupuncture will start on Day 0 and continue once daily to Day 15, as long as the patient is inpatient or comes to the clinic for post-transplantation follow-up. to prevent severe pain. If acupuncture does not prevent severe pain, the participant will receive opioid medication as backup pain relief.
  Acupuncture: Acupuncture treatments will be scheduled to cover the period of high symptom burden. Acupuncture will start on Day 0 and continue once daily to Day 15, as long as the patient is inpatient or comes to the clinic for post-transplantation follow-up. Electrical stimulation (e-acupuncture) may be applied to the ST36 and SP6 points when appropriate as per standard acupuncture practice.
  opioid: All study patients will receive the usual HSCT care and pain management regimens (usually opioids) as per standard practice at the study institution.
  Assessments: Participants will be asked to complete patient reported outcomes assessments online using REDCap or, If they prefer, via pencil and paper or over the phone. Assessments at baseline (within 4 weeks before HiChemo) and on or about days 7, 15, 30, and 90 after the first dose of HiChemo.
Period: Overall Study
Arm/Group | Acupuncture Plus Usual Care | Usual Care
Started | 151 | 147
Completed | 141 | 134
Not Completed | 10 | 13
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 8 | 10
Not completed — Disease progression | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture Plus Usual Care | Usual Care | Total
Number analyzed (Participants) | 151 | 147 | 298
Age, Continuous [Mean (Full Range); unit: years] | 58.4 [24.8 to 77.7] | 58.1 [19.2 to 75.3] | 58.3 [19.2 to 77.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 68 | 141
  Male | 78 | 79 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 141 | 135 | 276
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 10 | 7 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 20 | 15 | 35
  White | 114 | 121 | 235
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 151 | 147 | 298

OUTCOME MEASURES:

1. Primary Outcome: the Number of Patients Using Opioids at a Given Time
Description: at a given time divided by the total number of patients randomized to that group at Day 7) by review of medication records and urine drug test
Time Frame: at day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture Plus Usual Care | Usual Care
Number analyzed (Participants) | 141 | 134
Participants
  Using Opioid | 35 | 43
  No Opioid Use | 106 | 91

2. Primary Outcome: the Number of Patients Using Opioids at a Given Time
Description: at a given time divided by the total number of patients randomized to that group at Day 90) by review of medication records and urine drug test
Time Frame: at day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture Plus Usual Care | Usual Care
Number analyzed (Participants) | 141 | 134
Participants
  Using Opioid | 6 | 8
  No Opioid Use | 135 | 126

3. Primary Outcome: Symptom Burden
Description: measured by M. D. Anderson Symptom Inventory Blood and Marrow Transplantaion (MDASI-BMT). The symptoms rated are feeling physically sick, weak, diarrhea, mouth sores, and bleeding. All symptoms are rated with reference to "the last 24 hours" on 0-10 numeric scales from "not present" to "as bad as you can imagine." MDASIBMT Total Symptom Severity score will serve as the symptom burden primary endpoint. The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 numerical scale with 0 being "not present" and 10 being "as bad as you can imagine. Total symptom severity was calculated by averaging all 18 items in the scale
Time Frame: At baseline
Measure: Mean (95% Confidence Interval); unit: MDASIBMT Total Symptom Severity score
Arm/Group | Acupuncture Plus Usual Care | Usual Care
Number analyzed (Participants) | 141 | 134
MDASIBMT Total Symptom Severity score | 2.06 [1.86 to 2.25] | 2.06 [1.86 to 2.26]

4. Primary Outcome: Symptom Burden
Description: as for outcome 3
Time Frame: At Day 7
Measure: Mean (95% Confidence Interval); unit: MDASIBMT Total Symptom Severity score
Arm/Group | Acupuncture Plus Usual Care | Usual Care
Number analyzed (Participants) | 141 | 134
MDASIBMT Total Symptom Severity score | 2.96 [2.66 to 3.26] | 2.95 [2.63 to 3.27]

5. Primary Outcome: Symptom Burden
Description: as for outcome 3
Time Frame: At Day 90
Measure: Mean (95% Confidence Interval); unit: MDASIBMT Total Symptom Severity score
Arm/Group | Acupuncture Plus Usual Care | Usual Care
Number analyzed (Participants) | 141 | 134
MDASIBMT Total Symptom Severity score | 1.46 [1.20 to 1.72] | 1.40 [1.12 to 1.68]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Acupuncture Plus Usual Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/147
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/147
Other Adverse Events (participants affected / at risk) | 39/151 | 0/147
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acupuncture Plus Usual Care (N=151) | Usual Care (N=147)
Bruising (Injury, poisoning and procedural complications) | 26 | 0
Burning sensation (General disorders) | 1 | 0
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Foot cramping (Musculoskeletal and connective tissue disorders) | 1 | 0
Nose bleed (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pain/Soreness (General disorders) | 7 | 0
Throbbing sensation (General disorders) | 1 | 0
Tiredness (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04459416/Prot_SAP_000.pdf